CLINICAL TRIAL: NCT03081793
Title: Estimation of Average and Beat-to-beat Heart Rate With a Novel Wrist-worn PPG Device in Surgery Patients
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: PulseOn Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: Wristheartrate
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation
Keywords: postoperative monitoring; plethysmography; monitoring
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with sinus Rhythm: Patients with sinus rhythm at the beginning of monitoring
- Atrial fibrillation: Patients with atrial fibrillation at the beginning of monitoring

SUMMARY:
The aim of the study is to the reliability and feasibility of a novel optical heart rate monitor in hospital patients. Especially patients with atrial fibrillation are included. Patients will be monitored for two hours during routine post-operative care. The data from study device will be compared to routine monitoring. The design of the study is a Pilot feasibility study.

DETAILED DESCRIPTION:
The primary use of photoplethysmography (PPG) measurement in clinical settings is usually the determination of the blood oxygen saturation level of the patient. The same device often reports also an average pulse rate of the subject.

If the subject has low blood perfusion in the hands or suffers from acute atrial fibrillation, the determination of the pulse rate is challenging and therefore the readings provided by current technology are unreliable.

Optical heart rate monitors (OHR) have recently become popular in sports and wellness applications and their performance in healthy subjects having normal blood perfusion in the extremities is well studied and documented and good accuracy has been shown healthy subjects. The performance of wrist-worn OHR monitors in hospital patients, however, has not been extensively studied.

The aim of the study is to test novel wrist-worn photoplethysmographic (PPG) device in surgery patients and study its feasibility in detecting heart rate and beat to beat heart rate of patients having normal sinus rhythm or arrhythmia, such as atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years
* Subjected to surgery at Tampere University Hospital
* Spontaneously ventilating
* Volunteering for the study
* Able to give a written informed consent

Exclusion Criteria:

* Having a cardiac pacemaker
* Surgical operation performed in wrist area or any other reason that prevents placing the wrist-worn device in correct location
* Neurological disease (e.g. Parkinson's) possibly causing notable amount of shivering
* Non-Caucasian skin colour
* Inability to give an informed consent
* Denial of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to surgery requiring post-operative care. A heterogenous sample of patients with atrial fibrillation and patients with sinus rhytm
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Recognition of the rhythm | 2 hours
  To verify that average heart rate (HR) and beat-to-beat heart rate estimation is reliable also with hospital patients having either normal sinus rhythm, atrial fibrillation, or other arrhythmia

SECONDARY OUTCOMES:
quantification of estimation errors | 2 hours
  To quantify the estimation errors of aforementioned parameters by comparing them to reference values obtained from the ECG
identification of PPG morphology | 2 hours
  To quantify difference in morphological and other features calculated from the PPG signals collected from sinus-rhythm and AF patients

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No